CLINICAL TRIAL: NCT04939597
Title: A Phase 3 Randomized, Placebo-Controlled Trial Evaluating Memantine for Neurocognitive Protection in Children Undergoing Cranial Radiotherapy as Part of Treatment for Primary Central Nervous System Tumors
Brief Title: A Study to See if Memantine Protects the Brain During Radiation Therapy Treatment for a Brain Tumor
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ACCL2031; NCI-2020-07502 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCL2031 (Other: Children's Oncology Group); COG-ACCL2031 (Other: DCP); ACCL2031 (Other: CTEP); U01CA246568 (NIH); U24CA196173 (NIH); UG1CA189955 (NIH)
Record Dates: First submitted 2020-10-01; First posted 2021-06-25 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-10

CONDITIONS: Central Nervous System Carcinoma
MeSH Terms: interventions — Specimen Handling; Mental Status and Dementia Tests; Magnetic Resonance Spectroscopy; Memantine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (memantine hydrochloride) (Experimental): Patients receive memantine hydrochloride orally PO QD for week 1 and then BID for weeks 2-24 in the absence of disease progression or unacceptable toxicity. Patients also complete cognitive testing over 20-30 minutes at baseline, end of radiation therapy, and at 3, 6, 12, 24, and 48 months. Patients undergo MRI and may optionally undergo blood sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Cognitive Assessment; Procedure: Magnetic Resonance Imaging; Drug: Memantine Hydrochloride; Other: Questionnaire Administration
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO QD for week 1 and then BID for weeks 2-24 in the absence of disease progression or unacceptable toxicity. Patients also complete cognitive testing over 20-30 minutes at baseline, end of radiation therapy, and at 3, 6, 12, 24, and 48 months. Patients undergo MRI and may optionally undergo blood sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Cognitive Assessment; Procedure: Magnetic Resonance Imaging; Drug: Placebo Administration; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Cognitive Assessment — Complete cognitive testing
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Memantine Hydrochloride — Given PO
  Other Names: Ebixia; Namenda
  Arms: Arm I (memantine hydrochloride)
Drug: Placebo Administration — Given PO
  Arms: Arm II (placebo)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial compares memantine to placebo in treating patients with primary central nervous system tumors. Memantine may block receptors (parts of nerve cells) in the brain known to contribute to a decline in cognitive function. Giving memantine may make a difference in cognitive function (attention, memory, or other thought processes) in children and adolescents receiving brain radiation therapy to treat a primary central nervous system tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the efficacy, as measured by the slope of change of the Cogstate composite Z score from baseline to 12 months, of oral memantine hydrochloride (memantine) administered for a period of 6 months, when compared to placebo, in children ages 4-18 receiving cranial or craniospinal radiotherapy for primary central nervous system tumors.

EXPLORATORY OBJECTIVES:

I. To determine if memantine is associated with improved cognitive function as measured for participants in the optional Children's Oncology Group (COG) Standardized Battery at 12 months.

II. To determine if memantine is associated with change in cognitive function versus (vs.) placebo as measured by Cogstate composite score at end of radiation therapy (RT), 3 and 6 months.

III. To determine if memantine is associated with differences in cognitive function vs. placebo as measured by Cogstate composite score at 24 and 48 months for participants in the optional COG Standardized Battery.

IV. To correlate early cognitive changes (end of RT, 3, 6, 12 months Cogstate composite score) with late cognitive function (24 and 48 months Cogstate composite score).

V. To correlate COG Standardized Battery scores to Cogstate composite scores at 12, 24, and 48 months.

VI. To estimate the 36-month disease-free and overall survival (of primary brain tumor) after memantine treatment compared to placebo.

VII. To correlate changes in quantitative volumetric magnetic resonance imaging (MRI) measurements of critical brain regions with cognitive function over time.

VIII. To evaluate impact of memantine versus placebo on molecular biomarkers associated with cognitive decline after radiotherapy.

IX. To determine whether oral memantine, when compared to placebo, is associated with reduction in the incidence of decline of composite Cogstate score at 12 months in children ages 4-18 receiving cranial radiotherapy for primary central nervous system tumors.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive memantine hydrochloride orally (PO) once daily (QD) for week 1 and then twice daily (BID) for weeks 2-24 in the absence of disease progression or unacceptable toxicity. Patients also complete cognitive testing over 20-30 minutes at baseline, end of radiation therapy, and at 3, 6, 12, 24, and 48 months. Patients undergo MRI and may optionally undergo blood sample collection throughout the trial.

ARM II: Patients receive placebo PO QD for week 1 and then BID for weeks 2-24 in the absence of disease progression or unacceptable toxicity. Patients also complete cognitive testing over 20-30 minutes at baseline, end of radiation therapy, and at 3, 6, 12, 24, and 48 months. Patients undergo MRI and may optionally undergo blood sample collection throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* >= 4 and < 18 years at time of study entry
* Patients must weigh 15 kg or greater at time of study entry
* Primary central nervous system tumors that have not received prior cranial radiotherapy
* Planned focal, cranial or craniospinal radiation treatment for a primary central nervous system tumor
* The patient must have receptive and expressive language skills in English, French or Spanish since the neurocognitive function and quality of life (QOL) assessment instruments are available in these languages only
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or a serum creatinine based on age/sex as follows:

  * Age: 4 to < 6 years; Maximum serum creatinine (mg/dL): 0.8 male; 0.8 female
  * Age: 6 to < 10 years; Maximum serum creatinine (mg/dL): 1 male; 1 female
  * Age: 10 to < 13 years; Maximum serum creatinine (mg/dL): 1.2 male; 1.2 female
  * Age: 13 to < 16 years; Maximum serum creatinine (mg/dL): 1.5 male; 1.4 female
  * Age: >= 16 years; Maximum serum creatinine (mg/dL): 1.7 male; 1.4 female
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 135 U/L

  * Note: For the purpose of this study, the ULN for SGPT (ALT) has been set to the value of 45 U/L
* The patient must be able to undergo magnetic resonance imaging
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Life expectancy of less than 18 months
* Pre-existing conditions:

  * Any contraindication or allergy to study drug (memantine or placebo)
  * Intractable seizures while on adequate anticonvulsant therapy, defined as more than one seizure per month for the past 2 months or since initiating anticonvulsant therapy
  * History of neurodevelopmental disorder such as Down syndrome, Fragile X, William's Syndrome, intellectual disability (presumed intelligence quotient [IQ] < 70), etc
  * Co-morbid systemic illnesses, psychiatric conditions, social situations, or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens or would limit compliance with the study requirements
  * Patients with a motor, visual, or auditory condition that precludes participation in computerized neurocognitive assessments
  * Patients with any medical condition or taking medications that lead to alterations of urine pH towards the alkaline condition (e.g., renal tubular acidosis, carbonic anhydrase inhibitors, sodium bicarbonate)
* Personal history of prior cranial or craniospinal radiotherapy is not allowed

  * Note: Prior anti-cancer therapy including surgery, chemotherapy, targeted agents are allowed as per standard of care clinical treatment guidelines
* Female patients who are pregnant are excluded since fetal toxicities and teratogenic effects have been noted for the study drug. A pregnancy test is required for female patients of childbearing potential
* Lactating females who plan to breastfeed their infants
* Sexually active patients of reproductive potential who do not agree to use an effective contraceptive method for the duration of their study participation

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 192 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
The mean slope of the Cogstate composite Z score (an average of detection, Identification, and one-back Z scores, each Z score calculated using Cogstate age-based normative data) | Up-to 12 months post baseline
  We will estimate the difference in mean Cogstate composite Z score slopes (reflecting change in Cogstate composite Z scores from baseline to 12 months post baseline taking into account measurements at those time points as well as end of radiation therapy and 3 and 6-months post baseline between the treatment and control arms using a generalized estimating equation model with compound symmetry correlation structure and will provide a point estimate and corresponding 95% confidence interval.

OTHER OUTCOMES:
Intelligence quotient score (assessed by age-appropriate Wechsler Intelligence Scale) | At 12-months post baseline
  We will estimate the difference in mean standard scores across treatment arms and will provide a point estimate and corresponding 95% confidence interval.
Processing speed score (assessed by processing speed/attention subtests of age-appropriate Wechsler Intelligence Scale) | At 12-months post baseline
  We will estimate the difference in mean standard scores and will provide a point estimate and corresponding 95% confidence interval.
Verbal memory score (assessed by Children's Memory Scale [CMS] Stories subtest, or the Wechsler Memory Scale - Fourth Edition [WMS-IV] Logical Memory I and II subtests, depending on age) | At 12-months post baseline
  We will estimate the difference in mean standard scores across treatment arms and will provide a point estimate and corresponding 95% confidence interval.
Visual memory score (assessed by CMS or WMS-IV Faces subtest scores, Immediate and Delayed, depending on age) | At 12-months post baseline
  We will estimate the difference in mean standard scores across treatment arms and will provide a point estimate and corresponding 95% confidence interval.
Working memory score (assessed by Digit Span subtests of age-appropriate Wechsler Intelligence Scales) | At 12-months post baseline
  We will estimate the difference in mean standard scores across treatment arms and will provide a point estimate and corresponding 95% confidence interval.
Verbal score (assessed by the California Verbal Learning Test - Children's Version [CVLT-C] or 2nd Edition [CVLT-II] based on age, using the List A Trials 1-5 Total T-score) | At 12-months post baseline
  We will estimate the difference in mean standard scores and will provide a point estimate and corresponding 95% confidence interval.
Visual learning score (assessed by CMS Dot Locations subtest or WMS-IV Symbol Span subtest, depending on age) | At 12-months post baseline
  We will estimate the difference in mean standard scores across treatment arms and will provide a point estimate and corresponding 95% confidence interval.
Executive functioning score (assessed by the Cognitive Regulation Index of the Brief Rating Inventory of Executive Function) | At 12-months post baseline
  We will estimate the difference in mean standard scores across treatment arms and will provide a point estimate and corresponding 95% confidence interval.
Disease-free survival | Up-to 36 months post baseline
  We will estimate the hazard ratio comparing time-to-relapse of primary brain tumor or death due to any cause in the memantine relative to placebo arm and will provide a point estimate and corresponding 95% confidence interval.
Overall survival | Up-to 36 months post baseline
  We will estimate the hazard ratio comparing time-to- death due to any cause in the memantine relative to placebo arm and will provide a point estimate and corresponding 95% confidence interval.
Quantitative volumetric magnetic resonance imaging (MRI) measurements of critical brain regions (hippocampus, frontal cortex) | At 12-months post baseline
  We will estimate a correlation coefficient between changes in quantitative volumetric MRI measurements for the three regions of interest and changes in Cogstate composite Z scores (from baseline to 12 months post baseline).
Number of patients who consented to biobanking | Up-to 12 months post baseline
  The number of patients who agree to be in the biobanking part of the study future research.
Composite cognitive score decline (0.5 standard deviation or more decline in Cogstate composite score relative to baseline) | At 12-months post baseline
  We will estimate the proportion of patients who experience composite cognitive score decline in the memantine and placebo arms and will provide corresponding 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia N Laack, Principal Investigator — Children's Oncology Group
Locations (138):
- United States (137):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Maine Children's Cancer Program, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Albany Medical Center, Albany, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- HIMA San Pablo Oncologic Hospital, Caguas, Puerto Rico